CLINICAL TRIAL: NCT05354479
Title: Efficacy of Expressed Breast Milk Alone or in Combination With Paracetamol in Reducing Pain During ROP Screening
Brief Title: Breastmilk Alone or in Combination With Paracetamol for Reducing Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Rumpa Mani Chowdhury, DR, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 585
Record Dates: First submitted 2022-04-26; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Pain Control
MeSH Terms: conditions — Agnosia | interventions — Acetaminophen; Milk, Human

STUDY DESIGN:
Intervention Model Description: Double blinded Randomized control trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Both investigator and outcome assessor will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Expressed breast milk (Active Comparator): Babies will get only expressed breast milk.
  Interventions: Drug: Paracetamol
- paracetamol plus expressed breast milk (Experimental): Babies will get expressed breast milk plus paracetamol
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Drug: Paracetamol — babies will get expressed breast milk along with paracatamol for pain relief
  Other Names: Breast milk

SUMMARY:
Efficacy of Expressed Breast Milk Alone or in Combination with Paracetamol in Reducing Pain during ROP Screening.

DETAILED DESCRIPTION:
Retinopathy of prematurity (ROP) has been widely acknowledged to be the primary cause of preventable childhood blindness in developing countries. However, the procedure for screening is extremely painful. In this study, we will attempt to relieve the pain experienced by these babies using breast milk alone or in combination with oral paracetamol. This randomized control trial study will be conducted with the aim to assess the efficacy of Expressed Breast Milk Alone or in Combination with Paracetamol in Reducing Pain during ROP Screening. All preterm neonate who undergone ROP screening will be the study population. A total of 60 preterm neonates will be randomized into three groups: (Group A - control group = 20, Group B - breast milk group = 20, and Group C - oral paracetamol + breast milk = 20). Group A will get current care as per institutional protocol, Group B received 2 ml expressed breast milk (EBM) through a sterile syringe orally 2 min prior to procedure, Group C received syrup paracetamol, 15 mg/kg 30 min prior to procedure and EBM as in Group B. Pain experienced was measured by the premature infant pain profile (PIPP) score 20 s prior, during and 2 min after procedure. All procedures were video recorded. The Ophthalmologist and analyzer both will be blinded to the intervention. Results will be incorporated after enrollment

ELIGIBILITY:
Inclusion Criteria:

* 1. Gestational age <35 weeks, and birth weight <2000 gm

Exclusion Criteria:

* 1. Parents of neonate who refused to participate in the study 2. Newborns with multiple congenital anomalies 3. Patient who is on mechanical ventilator during ROP examination 4. Neonate receiving narcotic or sedative drugs 5. Neonate not receiving oral feed.

Ages: 20 Days to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-04-19 (Estimated); Study Completion 2022-04-19 (Estimated)

PRIMARY OUTCOMES:
Decrease in pain | 6 months
  Premature Infant Pain Score

CONTACTS AND LOCATIONS:
Locations (1):
- BSMMu, Dhaka, Bangladesh